CLINICAL TRIAL: NCT03940040
Title: Comparing the Effect of High Flow Nasal Oxygen With Usual Care on Pulmonary Rehabilitation in COPD Patients After an Acute Exacerbation; a Pilot Randomized Controlled Trial
Brief Title: High Flow Nasal Oxygen Versus Usual Care in COPD Pulmonary Rehabiliation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HFO_RCT
Record Dates: First submitted 2019-05-05; First posted 2019-05-07 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Patients will under go usual care ( pulmonary rehabilitation on room air or with nasal oxygen supplementation)
  Interventions: Other: Usual care
- High flow nasal oxygen (Experimental): Patients will undergo pulmonary rehabilitation with high flow nasal oxygen
  Interventions: Other: High flow nasal oxygen

INTERVENTIONS:
Other: Usual care — Usual Care
  Arms: Usual Care
Other: High flow nasal oxygen — High flow nasal oxygen
  Arms: High flow nasal oxygen

SUMMARY:
To compare the effects of high flow nasal oxygen with usual care during an outpatient 6-week pulmonary rehabilitation program after hospitalization for COPD exacerbation.

DETAILED DESCRIPTION:
This is a pilot randomized controlled trial to compare the effects of high flow nasal oxygen with usual care during an outpatient 6-week pulmonary rehabilitation program after hospitalization for COPD exacerbation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years and above
2. Known diagnosis of COPD based on history AND spirometry demonstrating post bronchodilator FEV1/FVC ratio <0.7
3. Currently admitted inpatient for an acute COPD exacerbation as the primary diagnosis
4. Fit to participate in exercise therapy as determined by both physician and physiotherapist
5. Has the mental capacity to follow instructions
6. Experience shortness of breath on exertion
7. Have decreased ability to carry out activities due to shortness of breath
8. Willing to participate in the exercise program

Exclusion Criteria:

1. Uncontrolled/ unstable medical conditions such as severe chronic heart failure that make exercise unsafe
2. Pulmonary disorder other than COPD
3. Physical conditions that preclude the ability to participate in exercise or may impair exercise performance.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-05-28 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
6-minute walk distance | 6 weeks
  It is the maximum distance walked in 6 minutes

SECONDARY OUTCOMES:
COPD Assessment Test score | 3 weeks, 6 weeks and 1 month after completion of program
  Chronic obstructive pulmonary disease assessment test (CAT) score
Hospital Anxiety Depression Scale | 3 weeks, 6 weeks and 1 month after completion of program
  This scale has 2 subscale scores of 1) Depression 2) Anxiety. Scores of 0-7 = Normal, 8-10 = Borderline, 11-21 = Abnormal
Respiratory function test | 3 weeks, 6 weeks and 1 month after completion of program
  It is a test of respiratory function
6-minute walk distance | 3 weeks and 1 month after completion of program
  It is the maximum distance walked in 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Yingjuan Mok, MBBS, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No